CLINICAL TRIAL: NCT04203004
Title: Hypothermic Oxygenated Perfusion With Cytokine Filtration in Clinical Liver Transplantation: a Randomised Controlled Trial
Brief Title: HOPE With Cytokine Filtration in Liver Transplantation (Cyto-HOPE)
Acronym: Cyto-HOPE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Papa Giovanni XXIII Hospital (Other)
Responsible Party: Principal Investigator, Stefania Camagni, MD, Principal Investigator, Papa Giovanni XXIII Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HOPE-2
Record Dates: First submitted 2019-12-16; First posted 2019-12-18 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Liver Transplantation; Post-Reperfusion Syndrome; Ischaemia-Reperfusion Injury; Early Allograft Dysfunction
Keywords: Hypothermic oxygenated perfusion (HOPE); Cytokine filtration; Liver transplantation
MeSH Terms: conditions — Reperfusion Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HOPE-CytoSorb (Experimental): Patients transplanted with livers preserved by HOPE with cytokine filtration by CytoSorb, a CE approved medical device for extracorporeal cytokine removal
  Interventions: Procedure: HOPE with cytokine filtration by CytoSorb
- HOPE-standard (No Intervention): Patients transplanted with livers preserved by HOPE without cytokine filtration

INTERVENTIONS:
Procedure: HOPE with cytokine filtration by CytoSorb — Cytokine filtration during HOPE
  Arms: HOPE-CytoSorb

SUMMARY:
Ischemia-reperfusion injury (IRI) is unavoidably typical of solid organ transplantation.

Post-reperfusion syndrome (PRS), characterized by hemodynamic instability at reperfusion of the implanted graft, is a possible complication of liver transplantation. For sure, IRI plays a fundamental role in the multifactorial pathogenesis of PRS.

IRI and PRS are associated with a higher risk of early allograft dysfunction (EAD) and, consequently, graft failure.

Liver grafts from both extended criteria donors (ECD) and donation after circulatory death (DCD) are particularly susceptible to IRI and, accordingly, are at higher risk of PRS, EAD and graft failure. Anyway, in the present scenario of organ shortage, such donors greatly contribute to enlarge the organ pool. So, various strategies have been developed for the purpose of a safer use of this kind of grafts. Among them, ex vivo hypothermic oxygenated perfusion (HOPE) reduces IRI and is beneficial for high-risk liver grafts.

The pathogenesis of IRI is an extremely complex downstream inflammation process, involving many different cytokines, chemokines and growth factors. In particular, tumor necrosis factor-alfa (TNF-alfa), interleukin-6 (IL-6), IL-8 and endothelin-1 (ET-1) are crucial in the development of IRI in liver transplantation.

In experimental models, cytokine filtration during ex vivo lung perfusion (EVLP) was proved to be safe and effective in reducing inflammatory response and, thus, pulmonary edema development.

Since

* in liver transplantation, IRI and PRS are associated with a higher risk of EAD and graft failure
* liver grafts from ECD and DCD are particularly susceptible to IRI and are at higher risk of PRS, EAD and graft failure
* HOPE of high-risk liver grafts reduces IRI
* in solid organ transplantation, various cytokines, chemokines and growth factors are involved in the pathogenesis of IRI
* in experimental models of EVLP, cytokine filtration was proved to reduce inflammatory response and subsequent organ damage,

our hypothesis is that cytokine filtration during HOPE of high-risk liver grafts may potentiate the beneficial effects of HOPE, further reducing IRI and, consequently, further decreasing the incidence of PRS and EAD.

So, the aim of this study is to verify the feasibility and safety of cytokine filtration during end-ischemic HOPE of liver grafts.

DETAILED DESCRIPTION:
This is a monocentric, pilot, randomized controlled study. Each eligible transplant candidate will be enrolled once an eligible graft has been allocated to him/her. Each enrolled patient will be randomized to either the experimental arm (HOPE-CytoSorb) or the control arm (HOPE-standard).

End-ischemic HOPE will be performed at our center after standard procurement of the graft at the donor hospital, static cold storage preservation during transport and back-table preparation. Dual HOPE, by portal continuous flow and arterial pulsatile flow, will be pressure controlled: portal pressure will be ≤5 mmHg and mean arterial pressure will be ≤30 mmHg. HOPE will be performed in an open system, so the graft will swim in the perfusate flowing out of the vena cava. The recirculating perfusion solution will have the same composition of University of Wisconsin Machine Perfusion Solution. HOPE will be maintained for 4 hours. CytoSorb will be included in the circuit only in the experimental arm.

Scheduled samples of both the perfusate and patient's blood will be analyzed for the levels of TNF-alfa, IL-6, IL-8 and ET-1. A biopsy of the implanted graft will be taken 2 hours after its reperfusion. The patient will be followed for 1 year after transplantation.

Once 10 patients have been enrolled, an interim analysis will be performed by an independent Clinical Endpoint Committee.

ELIGIBILITY:
RECIPIENTS

* Inclusion criteria: age ≥18 years, signed informed consent form
* Exclusion criteria: age <18 years, combined liver-other organ transplantation, pre-transplant treatment with plasmapheresis, refusal to consent to the study

GRAFTS ELIGIBILITY CRITERIA TO HOPE:

* grafts from extended criteria donors with any combination of the following characteristics: age ≥70 years; macrosteatosis ≥35%; diabetes mellitus; severe vasculopathy; anti-HCV or HBsAg positivity (upon biopsy)
* grafts from donors with hemodynamic instability
* graft from DCD (occasionally)
* grafts with an anticipated long cold ischemia time
* PARTIAL GRAFTS ARE EXCLUDED FROM THE STUDY

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-09-23 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of post-reperfusion syndrome | Intraoperatively, during the first 5 minutes after reperfusion of the liver graft
  Aggarwal definition: a decrease in mean arterial pressure >30% below the baseline value, for at least 1 minute, occurring during the first 5 minutes after reperfusion of the liver graft

SECONDARY OUTCOMES:
Entity of ischemia-reperfusion injury | 2 hours after reperfusion of the liver graft
  Assessment of liver biopsy according to Suzuki histological grading system modified by UCLA group [Sosa RA et al. JCI Insight 2016; 1(20): e89679]
Incidence of early allograft dysfunction | Postoperative day 7
  Olthoff definition: presence of almost one of the following variables: bilirubin ≥10 mg/dl on postoperative day 7, INR ≥1.6 on postoperative day 7, ALT or AST >2000 UI/ml within the first 7 postoperative days

CONTACTS AND LOCATIONS:
Overall Officials: Michele Colledan, MD, FEBS, Study Director — Papa Giovanni XXIII Hospital
Locations (1):
- Papa Giovanni XXIII Hospital, Bergamo, Italy